CLINICAL TRIAL: NCT03812718
Title: Anaesthesia Requirements for Ventilation With Endotracheal Tube Versus ProSeal Laryngeal Mask Airway During Automated Feedback-Loop Controlled Total Intravenous Anaesthesia in Patients Undergoing Laparoscopic Cholecystectomy: A Randomised Controlled Study
Brief Title: Comparison of Anaesthesia Requirement for Ventilation With Endotracheal Tube Versus Proseal Laryngeal Mask Airway
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sir Ganga Ram Hospital (Other)
Responsible Party: Principal Investigator, Nitin Sethi, DNB, Consultant & Associate Professor, Sir Ganga Ram Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: EC/01/19/1464
Record Dates: First submitted 2019-01-19; First posted 2019-01-23 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Cholelithiases; Cholecystolithiasis
MeSH Terms: conditions — Cholelithiasis; Cholecystolithiasis

STUDY DESIGN:
Intervention Model Description: 160-patients will be randomly divided into one of the two groups:
  Group-I (ETT group, n= 80) ETT will be used as the airway device for maintaining ventilation
  Group-2 (PLMA group, n= 80) PLMA will be used as the airway device for maintaining ventilation
Who Masked: Participant, Outcomes Assessor
Masking Description: The attending anaesthesiologist will not be blinded to the technique utilized to administer GA. An independent assessor unaware of the technique utilized for administering GA will analyse the intraoperative data and conduct the postoperative follow up
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ETT Group (Active Comparator): Anesthesia will be induced with fentanyl-citrate (3µg/kg) and propofol (dose determined by automated system based on continuous BIS feedback from the patients). Atracurium besylate 0.5-mg/kg will be given to facilitate placement of airway device. Propofol administration rate will be controlled by a feedback loop facilitated by BIS monitoring using the closed-loop anaesthesia delivery system (CLADS). A BIS value of 50 will be used as the target point for induction and maintenance of GA.
  Intraoperative ventilation will be instituted through a polyvinyl chloride (PVC) ETT (Portex, Smiths Medical ASD, Inc, Minneapolis, USA). The size of the tube will be standardized for the male (7.5 mm ID) and the female (6.5 MM ID).
  Interventions: Device: Endotracheal tube (ETT)
- PLMA Group (Active Comparator): Anesthesia will be induced with fentanyl-citrate (3µg/kg) and propofol (dose determined by automated system based on continuous BIS feedback from the patients). Atracurium besylate 0.5-mg/kg will be given to facilitate placement of airway device. Propofol administration rate will be controlled by a feedback loop facilitated by BIS monitoring using the closed-loop anaesthesia delivery system (CLADS). A BIS value of 50 will be used as the target point for induction and maintenance of GA. intraoperative ventilation will be maintained with PLMA (Telefex Medical, Westmeath Ireland) whose size would be selected based on body weight. In patients weighing 30-50 kg PLMA # 3.0, 50-70 kg PLMA # 4.0, and 50-100 kg PLMA # 5.0 will be inserted.
  Interventions: Device: ProSeal Laryngeal Mask Airway (PLMA)

INTERVENTIONS:
Device: Endotracheal tube (ETT) — After induction of anaesthesia patient will be intubated with polyvinyl chloride (PVC) ETT for maintaining intraoperative ventilation. Anaesthesia will be maintained with propofol and the administration rate will be controlled by a feedback loop facilitated by BIS monitoring using the closed-loop anaesthesia delivery system (CLADS). A BIS value of 50 will be used as the target point for induction and maintenance of GA.
  Arms: ETT Group
Device: ProSeal Laryngeal Mask Airway (PLMA) — After induction of anaesthesia ProSeal Laryngeal Mask Airway (PLMA) will be inserted for maintaining intraoperative ventilation. Anaesthesia will be maintained with propofol and the administration rate will be controlled by a feedback loop facilitated by BIS monitoring using the closed-loop anaesthesia delivery system (CLADS). A BIS value of 50 will be used as the target point for induction and maintenance of GA.
  Arms: PLMA Group

SUMMARY:
Endotracheal tube (ETT) is the gold standard conduit for providing controlled ventilation during general anaesthesia (GA). however, the supra-glottic airway (SGA) devices in particular the laryngeal mask airway (LMA) and its variants have become a reliable alternative to ETT for carrying out controlled ventilation. Of the several variants of LMA available today, the proseal LMA (PLMA) is preferred for controlled ventilation. The various advantages of LMA includes, a lower incidence of postoperative sore throat and superior haemodynamic profile during surgery. However, one aspect of providing anaesthesia with LMA compared to ETT is the ability of LMA to maintain equivalent depth of anaesthesia with lower anaesthetic requirement, is quiet intriguing and evidence to this regard is very limited.

By measuring the anaesthesia requirement using a robust computerised delivery system such as the closed loop anaesthesia delivery system (CLADS) we can establish for sure the anaesthesia required for maintaining intraoperative mechanical ventilation with the use of these two (ETT and PLMA) airway management devices.

This randomised controlled study aims to calculate the anaesthesia requirement as determined by the total amount of propofol consumed for maintaining anaesthesia with ETT versus PLMA

DETAILED DESCRIPTION:
Endotracheal tube (ETT) is the gold standard conduit for providing controlled ventilation during general anesthesia (GA). However, since the introduction of classic laryngeal mask airway (LMA) in the 1980's and serial evolution of supra-glottic airway devices (SGA) thereafter, LMAs have become a reliable alternative to ETT for carrying out controlled ventilation. Interestingly, of the additional advantages that the LMA proffers, including, a lower incidence of postoperative sore throat (POST) and superior hemodyamic profile during surgery; its ability to maintain equivalent depth of anesthesia (in comparison to when ETT-GA) with lower anesthetic requirement, is intriguing.

A handful of studies have demonstrated that the end-tidal isoflurane concentration required for maintenance of GA is 0.2 -0.53% greater with use of ETT as compared to LMA. However, the evidence generated by these studies remains unsubstantiated because in them, anaesthetic gas concentration was titrated to patient's clinical profile like heart rate and blood pressure without the backing of specific protocol for maintaining depth-of-anaesthesia. Therefore, for credible evidence, assessment of quantitative anesthetic requirement for achieving and sustaining a steady anesthesia depth with either LMA or ETT warrants confirmation with the use of an objective depth-of-anesthesia monitor, such as, bispectral index (BIS).

Closed loop anaesthesia delivery system (CLADS) is an indigenously developed patented (502/DEL/2003) computer-controlled and BIS-guided automated anesthesia delivery system. CLADS, which runs on a control algorithm based on the relationship between diverse rates of propofol infusion and the processed EEG variable; delivers propofol infusion at a rate which is continuously adjusted by patient's state of depth of anesthesia as per BIS monitoring input. This automated system maintains anaesthesia depth with high accuracy and objectively determines propofol delivery quantitatively.

Of the several variants of SGA available today, the ProSeal laryngeal mask airway (PLMA) 9 is preferred for controlled ventilation for its unique design that serves dual function of a ventilation tube and an oropharyngeal drainage tube for excluding gastric contents from getting aspirated through the peri-laryngeal cuff seal.

Given that CLADS can help us to accurately quantify anaesthesia, we hypothesize that there is no difference in anesthesia requirement for GA maintained through an ETT or a PLMA. This randomized controlled study aims to compare: anaesthesia requirement as determined by total propofol consumption (primary objective); intraoperative hemodynamic profile and incidence of POST (secondary objectives) in patients undergoing laparoscopic surgery with controlled ventilation via ETT or PLMA.

ELIGIBILITY:
Inclusion Criteria:

1. ASA physical status I/II
2. Undergoing elective laparoscopic cholecystectomy

Exclusion Criteria:

1. Anticipated difficult airway
2. Body mass index > 30-kg/m2
3. Uncompensated cardiovascular disease (e.g. uncontrolled hypertension, atrio-ventricular block, sinus bradycardia, congenital heart disease, reduced LV compliance, diastolic dysfunction)
4. Hepato-renal insufficiency
5. Uncontrolled endocrinology disease (e.g. diabetes mellitus, hypothyroidism)
6. Known allergy/hypersensitivity to the study drug (propofol)
7. Drug dependence/substance abuse/psychiatric illness
8. Requirement of postoperative ventilation
9. Refusal to informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2019-03-04 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in Propofol usage in milligrams | From beginning of anaesthesia (0-hours, baseline) till 4 hours intraoperatively
  Comparison of quantitative difference in propofol requirement between the two groups

SECONDARY OUTCOMES:
Anaesthesia depth consistency using BIS scores | From beginning of anaesthesia (0-hours, baseline) till 3 hours intraoperatively
  Determined by the percentage of the total anaesthesia time in which the BIS scores remain within a score of 10% of the target BIS (i.e. BIS-50) in both the study arms.
Evaluation of propofol anaesthesia delivery system | From beginning of anaesthesia (0-hours, baseline) till 3 hours intraoperatively
  Determined by using Varvel criteria parameters; median performance error (MDP), median absolute performance error (MDAPE), wobble and global score in both the study arms
Change in Intra-operative heart Rate (beats per minute) | From beginning of anaesthesia (0-hours, baseline) till 3 hours intraoperatively
  Comparison of intra-operative heart rate between both the arms will be done
Change in Intra-operative systolic , diastolic, and mean (mmHg) | From beginning of anaesthesia (0-hours, baseline) till 10 hours intraoperatively
  Comparison of intra-operative blood pressure- systolic, diastolic, and mean between both the arms will be done
Early Recovery from anesthesia | From end of anaesthesia till 20-minutes postoperatively
  Time taken by the patient to open his/her eyes after discontinuation of anaesthesia will be noted
Post operative sedation | From the end of anaesthesia till 24-hours, postoperatively
  Will be assessed using Modified Observer's assessment of alertness/sedation scale (MOAA/S)
Incidence of postoperative sore throat | From the end of anaesthesia till 24-hours, postoperatively
  Comparison of post operative sore throat occurrence between the two groups

CONTACTS AND LOCATIONS:
Overall Officials: Nitin Sethi, DNB, Principal Investigator — Sir Ganga Ram Hospital; Amitabh Dutta, MD, Study Director — Sir Ganga Ram Hospital; Jayashree Sood, MD, FFRCA, Study Chair — Sir Ganga Ram Hospital
Locations (1):
- Sir Ganga Ram Hospital, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No